Official Title: Communicating Waterpipe Tobacco Harms to Reduce Use Among Young Adults: Aim 2

Text Versus Pictorial Warning Survey

NCT05783843

IRB-Approved Date: 1/27/23

WTW Aim 2 TVPS – Consent CLEAN 1/26/2023

## Consent

## Creating Waterpipe Tobacco Warnings to Reduce Use among Young Adults Aim 2: Text v. Pictorial Warning Survey

## Wake Forest Health Survey

You are invited to complete a survey as part of a research study being conducted by Wake Forest School of Medicine. The goal of the survey is to understand what young adults think about different examples of hookah tobacco packages. You will be shown up to six packages and will answer questions about each one. The survey will take about 15 minutes to complete. We expect that about 1,200 people will complete the survey. There is no cost to you to take the survey. Upon completion of the survey, you will be provided with compensation agreed upon with your panel. Your participation is completely voluntary. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. You may choose not to take part or you may leave the study at any time.

The risk of harm or discomfort that may happen as result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. There is a slight risk of breach of confidentiality. We will do our best to protect your confidential information. Efforts, such as coding research records, keeping research records secure, and only allowing authorized people to have access to research records will be made to keep your information safe. No reference to any individual participant will appear in reports, presentations, or publications that may arise from the study. Identifiers might be removed from the identifiable private information and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future. This study is not intended to provide treatment for any disease or condition. The alternative to participating in the study is to not participate.. The person in charge of this study is Erin Sutfin, PhD. If you have any questions, suggestions, or concerns regarding this survey, or if you wish to withdraw from the study, please contact Dr. Sutfin at <a href="https://hookahresearch@wakehealth.edu">hookahresearch@wakehealth.edu</a>. If you have any questions, suggestions, or concerns about your rights as a volunteer in this research, please contact the Wake Forest Institutional Review Board at Wake Forest Research Subject Advocate at The Concerns and the Concerns and the Concerns are contact the Wake Forest Institutional Review Board at The Concerns and the Concerns are contact the Wake Forest Research Subject Advocate at The Concerns are contact the Wake Forest Research Subject Research Subje

Checking the box below indicates that:

- You have read the above information and have had a chance to ask questions about being in this study and having those questions answered
- You voluntarily agree to participate
- You are at least 18 years of age
- You authorize the use and disclosure of your health information as described in this consent and authorization form
- You understand that by taking part in this study, you are not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence

| Chack "I | agroo" | if you wo | ıld lika t | o participate | |
|----------|--------|------------|------------|---------------|---|
| Cneck I | auree | ıı vou wol | lia iike i | o participate | _ |

| I agree |
|----------------|
| I do not agree |